CLINICAL TRIAL: NCT03751813
Title: Baby Bump Lifestyle Intervention Supplement Study
Acronym: Baby BLISS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB had concerns about study; terminated
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Kai Ling Kong, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Baby BLISS
Record Dates: First submitted 2018-11-19; First posted 2018-11-23 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): placebo supplement
  Interventions: Dietary Supplement: Supplement
- Supplement (Experimental): actual supplement
  Interventions: Dietary Supplement: Supplement

INTERVENTIONS:
Dietary Supplement: Supplement — Supplement will be given to this group to take daily for 8 weeks

SUMMARY:
The overall purpose of this study is to examine how natural supplements can mediate the effects of stress on fetal development during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman presenting to her first obstetrical visit for this pregnancy
* Must be in the first trimester (<13 weeks)
* 18 years or older
* High-stress levels as measured by the Perceived Stress Level Questionnaire
* Must be a single pregnancy (e.g. not twins, triplets, etc.)

Exclusion Criteria:

* Diabetes (types 1 and 2)
* Diagnosis of gestational diabetes in prior pregnancy
* Hyperemesis gravidarum or severe morning sickness that interferes with supplement intake
* Major medical illnesses including but not limited to: malabsorption syndromes (Celiac's disease, Crohn's, Ulcerative Colitis), Systemic Lupus Erythematosus and other major autoimmune conditions

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 4 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
lower blood stress markers via venous draw | 9 months
  We hypothesize that the addition of nutrients during gestation will decrease the levels of stress hormones/reactants in pregnant women who are at high risk for stressful pregnancies.

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No